CLINICAL TRIAL: NCT01297517
Title: Three Month Efficacy and Safety Study of a Fixed Combination of Brinzolamide 1%/Brimonidine 0.2% Compared to Brinzolamide 1% and Brimonidine 0.2% All Dosed Three Times Daily in Patients With Open-Angle Glaucoma and/or Ocular Hypertension
Brief Title: Efficacy and Safety Study of Brinzolamide 1%/Brimonidine 0.2% vs. Brinzolamide 1% and Brimonidine 0.2%
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C-10-033
Record Dates: First submitted 2011-02-15; First posted 2011-02-16 (Estimated); Results first posted 2013-05-13 (Estimated); Last update posted 2013-05-21 (Estimated); Status verified 2013-05

CONDITIONS: Open-Angle Glaucoma; Ocular Hypertension
Keywords: AOG; OHT; Open-Angle Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — brinzolamide; Brimonidine Tartrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Brinzolamide/Brimonidine (Experimental): Brinzolamide 1%/brimonidine tartrate 0.2% ophthalmic suspension, one drop instilled in each eye three times a day for 3 months
  Interventions: Drug: Brinzolamide 1%/brimonidine tartrate 0.2% ophthalmic suspension
- Brinzolamide (Active Comparator): Brinzolamide ophthalmic suspension, 1%, one drop instilled in each eye three times a day for 3 months
  Interventions: Drug: Brinzolamide ophthalmic suspension, 1%
- Brimonidine (Active Comparator): Brimonidine tartrate ophthalmic solution, 0.2%, one drop instilled in each eye three times a day for 3 months
  Interventions: Drug: Brimonidine tartrate ophthalmic solution, 0.2%

INTERVENTIONS:
Drug: Brinzolamide 1%/brimonidine tartrate 0.2% ophthalmic suspension
  Arms: Brinzolamide/Brimonidine
Drug: Brinzolamide ophthalmic suspension, 1%
  Other Names: AZOPT®
  Arms: Brinzolamide
Drug: Brimonidine tartrate ophthalmic solution, 0.2%
  Arms: Brimonidine

SUMMARY:
The purpose of this study was to evaluate the efficacy and safety of a fixed combination of Brinzolamide/Brimonidine in lowering intraocular pressure (IOP) relative to each of its individual active components in patients with open-angle glaucoma and/or ocular hypertension.

DETAILED DESCRIPTION:
This study consisted of 6 visits conducted during 2 sequential phases: the Screening/Eligibility phase, which included a screening visit and 2 eligibility visits, and the Treatment phase, which included 3 on-therapy visits conducted at Week 2, Week 6, and Month 3. A washout period based on previous ocular medication preceded Eligibility Visit 1. Patients who met all inclusion/exclusion criteria at both eligibility visits were randomized (1:1:1) to receive treatment with 1 of 3 study drugs for 3 months. Study drug instillation began the morning after the second eligibility visit.

ELIGIBILITY:
Inclusion Criteria:

* Sign Informed Consent document.
* Diagnosis of open-angle glaucoma or ocular hypertension, with mean intraocular pressure within protocol-specified range at eligibility visit/s.
* Other protocol-specified inclusion criteria may apply.

Exclusion Criteria:

* Females of childbearing potential if pregnant, lactating, or not using highly effective birth control measures.
* Any form of glaucoma other than open-angle glaucoma.
* Severe central vision loss in either eye.
* Chronic, recurrent, or severe inflammatory eye disease.
* Ocular trauma within the preceding 6 months.
* Ocular infection or ocular inflammation within the preceding 3 months.
* Clinically significant or progressive retinal disease such as retinal degeneration, diabetic retinopathy, or retinal detachment.
* Best-corrected visual acuity score worse than 55 letters using the Early Treatment Diabetic Retinopathy Study chart.
* Other ocular pathology (including severe dry eye) that may, in the opinion of the Investigator, preclude the administration of study product.
* Ocular surgery within the preceding 6 months.
* Ocular laser surgery within the preceding 3 months.
* Any abnormality preventing reliable applanation tonometry.
* Any other conditions, including severe illness, which could make the patient, in the opinion of the Investigator, unsuitable for the study.
* Other protocol-specified exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1001 (Actual)
Dates: Start 2011-02; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Teague, BS, Sr. Clinical Manager, Study Director — Alcon Research

REFERENCES:
- [Derived] Katz G, Dubiner H, Samples J, Vold S, Sall K. Three-month randomized trial of fixed-combination brinzolamide, 1%, and brimonidine, 0.2%. JAMA Ophthalmol. 2013 Jun;131(6):724-30. doi: 10.1001/jamaophthalmol.2013.188. PMID 23579344

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 68 study centers in the US.
Pre-assignment Details: Of the 1001 enrolled, 341 subjects did not qualify for treatment and were exited without exposure to product. The 660 subjects eligible for treatment were randomized (1:1:1) to study drug. This reporting group includes all randomized subjects, as treated.
Groups:
- Brinzolamide/Brimonidine: Brinzolamide 1%/brimonidine tartrate 0.2% ophthalmic suspension, one drop instilled in each eye three times a day (8 am, 3 pm, 10 pm) for three months
- Brinzolamide: Brinzolamide ophthalmic suspension, 1%, one drop instilled in each eye three times a day (8 am, 3 pm, 10 pm) for three months
- Brimonidine: Brimonidine tartrate ophthalmic solution, 0.2%, one drop instilled in each eye three times a day (8 am, 3 pm, 10 pm) for three months
Period: Overall Study
Arm/Group | Brinzolamide/Brimonidine | Brinzolamide | Brimonidine
Started | 214 | 226 | 220
Completed | 187 | 214 | 193
Not Completed | 27 | 12 | 27
Not completed — Adverse Event | 21 | 7 | 16
Not completed — Lost to Follow-up | 1 | 0 | 1
Not completed — Patient Decision Unrelated to AE | 2 | 3 | 7
Not completed — Noncompliance | 1 | 0 | 0
Not completed — Protocol Violation | 1 | 1 | 1
Not completed — Inadequate Control of IOP | 1 | 1 | 2

BASELINE CHARACTERISTICS:
Population: This reporting group includes all participants randomized to study drug, as treated.
Groups:
- Total: Total of all reporting groups
Arm/Group | Brinzolamide/Brimonidine | Brinzolamide | Brimonidine | Total
Number analyzed (Participants) | 214 | 226 | 220 | 660
Age, Customized [Number; unit: participants]
  18 to 64 years | 107 | 101 | 117 | 325
  ≥65 years | 107 | 125 | 103 | 335
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 140 | 128 | 135 | 403
  Male | 74 | 98 | 85 | 257

OUTCOME MEASURES:

1. Primary Outcome: Mean IOP at Month 3 for Each Assessment Timepoint (8 AM, + 2 h, + 7 h, and + 9 h)
Description: At the Month 3 (Exit) visit, the 8 am IOP measurement was taken before instillation of study drug. The study drug was instilled approximately 15 minutes after the 8 am measurement. An additional dose was given at 3 pm. Intraocular pressure was measured by Goldmann applanation tonometry. One eye from each patient was chosen as the study eye and only data for the study eye were used for the efficacy analysis. A higher IOP can be a greater risk factor for developing glaucoma or glaucoma progression (leading to optic nerve damage).
Time Frame: Month 3
Population: Intent-to-treat (ITT): All patients who received study medication and completed at least 1 scheduled on-therapy study visit. Observed case analysis of the ITT dataset, per randomized treatment assignment.
Measure: Least Squares Mean (Standard Error); unit: millimeters mercury (mm Hg)
Arm/Group | Brinzolamide/Brimonidine | Brinzolamide | Brimonidine
Number analyzed (Participants) | 189 | 213 | 192
millimeters mercury (mm Hg)
  8 am (before study drug instillation) | 20.5 (0.29) | 21.6 (0.28) | 23.3 (0.29)
  +2 hrs relative to 8 am dosing | 17.2 (0.29) | 20.4 (0.28) | 19.7 (0.29)
  +7 hrs relative to 8 am dosing | 18.7 (0.29) | 20.4 (0.28) | 21.3 (0.29)
  +9 hrs relative to 8 am dosing | 17.0 (0.29) | 20.0 (0.28) | 18.8 (0.29)

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of the study (1 year). An AE was any untoward medical occurrence in a patient administered a study medication, regardless of whether or not the event had a causal relationship with the medication.
Description: This reporting group includes all participants randomized to study drug, as treated. Adverse events were obtained as solicited comments from the study patients and as observations by the study investigator as outlined in the study protocol.
Arm/Group | Brinzolamide/Brimonidine | Brinzolamide | Brimonidine
Serious Adverse Events (participants affected / at risk) | 2/214 | 6/226 | 2/220
Other Adverse Events (participants affected / at risk) | 20/214 | 26/226 | 1/220
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Brinzolamide/Brimonidine (N=214) | Brinzolamide (N=226) | Brimonidine (N=220)
Cardiac pacemaker insertion (Surgical and medical procedures) | 1 | 0 | 0 — Not related
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 — Not related
Chest pain (General disorders) | 0 | 1 | 0 — Related
Amnesia (Nervous system disorders) | 0 | 1 | 0 — Not related
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 — Not related
Angina pectoris (Cardiac disorders) | 0 | 1 | 0 — Not related
Collapse of lung (Injury, poisoning and procedural complications) | 0 | 1 | 0 — Not related
Vertebroplasty (Surgical and medical procedures) | 0 | 1 | 0 — Not related
Vulval neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 — Not related
Chest pain (General disorders) | 0 | 0 | 2 — Not related
Injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 — Not related
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Brinzolamide/Brimonidine (N=214) | Brinzolamide (N=226) | Brimonidine (N=220)
Vision blurred (Eye disorders) | 14 | 15 | 1
Dysgeusia (Nervous system disorders) | 8 | 14 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.